CLINICAL TRIAL: NCT01307020
Title: Double-blind, Randomised, Placebo and Active Controlled, Parallel Group Study to Evaluate the Analgesic Effect of a Single Oral Administration of Four Different Combination Doses of DKP.TRIS With TRAM.HCL in Comparison With the Single Agents, on Moderate to Severe Pain Following Impacted Third Mandibular Molar Tooth Extraction
Brief Title: Analgesic Effect of Different Combinations of Dexketoprofen Trometamol With Tramadol Hydrochloride in a Model of Moderate to Severe Pain
Acronym: DEX-TRA 02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEX-TRA 02; 2010-022798-32 (EudraCT Number)
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-07

CONDITIONS: Pain
Keywords: Moderate to severe pain; Postoperative pain; Analgesics; Dexketoprofen; Tramadol
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — dexketoprofen trometamol; Tramadol; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- TRAM.HCl high dose (Active Comparator)
  Interventions: Drug: Tramadol Hydrochloride
- TRAM.HCl low dose (Active Comparator)
  Interventions: Drug: Tramadol Hydrochloride
- DKP-TRIS high dose (Active Comparator)
  Interventions: Drug: Dexketoprofen Trometamol
- DKP-TRIS low dose (Active Comparator)
  Interventions: Drug: Dexketoprofen Trometamol
- DKP-TRIS low dose - TRAM.HCl low dose (Experimental)
  Interventions: Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride
- DKP-TRIS low dose - TRAM.HCl high dose (Experimental)
  Interventions: Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride
- DKP-TRIS high dose - TRAM.HCl low dose (Experimental)
  Interventions: Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride
- DKP-TRIS high dose - TRAM.HCl high dose (Experimental)
  Interventions: Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride

INTERVENTIONS:
Drug: Dexketoprofen Trometamol — Dexketoprofen Trometamol low dose, oral film-coated table, once
  Arms: DKP-TRIS low dose
Drug: Dexketoprofen Trometamol — Dexketoprofen Trometamol high dose, oral film-coated table, once
  Arms: DKP-TRIS high dose
Drug: Tramadol Hydrochloride — Tramadol Hydrochloride low dose, oral film-coated table, once
  Arms: TRAM.HCl low dose
Drug: Tramadol Hydrochloride — Tramadol Hydrochloride high dose, oral film-coated table, once
  Arms: TRAM.HCl high dose
Drug: Ibuprofen — Ibuprofen 400 mg, oral film-coated table, once
  Arms: Ibuprofen
Drug: Placebo — Placebo, oral film-coated table, once
  Arms: Placebo
Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride — DKP-TRIS low dose - TRAM.HCl low dose, oral film-coated table, once
  Arms: DKP-TRIS low dose - TRAM.HCl low dose
Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride — DKP-TRIS low dose - TRAM.HCl high dose, oral film-coated table, once
  Arms: DKP-TRIS low dose - TRAM.HCl high dose
Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride — DKP-TRIS high dose - TRAM.HCl low dose, oral film-coated tablet, once
  Arms: DKP-TRIS high dose - TRAM.HCl low dose
Drug: Dexketoprofen Trometamol + Tramadol Hydrochloride — DKP-TRIS high dose - TRAM.HCl high dose, oral film-coated tablet, once
  Arms: DKP-TRIS high dose - TRAM.HCl high dose

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy of Dexketoprofen Trometamol and Tramadol Hydrochloride given in combinations and the analgesic efficacy of each single component in comparison to placebo on moderate to severe pain following impacted third mandibular molar tooth extraction. Ibuprofen will be used as an active control to validate the pain model.

DETAILED DESCRIPTION:
The aim of this study is to develop a combination of Dexketoprofen Trometamol (DKP.TRIS) and Tramadol Hydrochloride (TRAM.HCl) for the treatment of acute moderate to severe pain, based on the rationale that more than one drug is necessary in most patients suffering of acute and chronic pain, particularly of moderate to severe intensity.

DKP.TRIS and TRAM.HCl have different mechanisms of action, therefore their combination is expect to result in an additive or synergistic analgesia, thus allowing a decrease in the required doses of the individual agents, and consequently a reduced risk of adverse events In this study, patients who present moderate to severe pain after impacted third mandibular molar tooth extraction will be randomised to a total of 10 treatment arms including 4 combinations of DKP.TRIS + TRAM.HCl, the four corresponding single treatments, placebo and ibuprofen. Treatment administration will be followed by a 24-hour pain and analgesic effect assessment.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting ALL the following criteria will be eligible for entry into the study:

* Male or female patients aged 18 to 70 years old. Females participating in the study must be either: of non-childbearing potential, or willing to use a highly effective contraceptive method.
* Scheduled for outpatient surgical extraction -under local anaesthesia- of third mandibular molar teeth, with at least one of which is fully or partially impacted in the mandible requiring bone manipulation.
* Normal physical examination or without clinically relevant abnormalities.

At randomisation (after surgery):

No intake of analgesics (including prescription and over the counter drugs) within 24h prior to the surgery.

* No complication during the surgery, duration of surgery < 1 hour and not requiring re-anaesthesia.
* Patients experiencing pain of moderate or higher intensity in the first four hours after the end of surgery.

Exclusion Criteria:

* History of allergy or hypersensitivity to NSAIDs, opioids or acetyl salicylic acid.
* History of asthma, bronchospasm, acute rhinitis, nasal polyps, urticaria or angioneurotic oedema.
* History of peptic ulcer, gastrointestinal disorders by NSAIDs, gastrointestinal bleeding or other active bleedings.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 745 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cosme Gay-Escoda, Professor, Study Chair — Department of Oral and Maxillofacial Surgery, School of Dentistry, University of Barcelona - Bellvitge Institute for Biomedical Research (IDIBELL) 08907 Hospitalet de Llobregat, Barcelona (Spain); R Andrew Moore, Professor, Study Chair — Pain Research & Nuffield Division of Anaesthesics, Department of Clinical Neurosciences, University of Oxford. The Churchill, Oxford OX3 7LJ (United Kingdom)
Locations (16):
- Germany (2):
  - Klinik und Polickinik für Mund-Kiefer-Gesichtschirurgie/Plastische Operationen Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Klinik für Mund-, Kiefer- und Gesichtschirurgie, Universitätsklinikum Schleswig Holstein, Campus Kiel, Kiel, Schleswig-Holstein
- Dr Tóth Bagi Zoltán Fogászati Rendeloje, Budapest, Budapest, Hungary
- Italy (2):
  - Centro di Farmacologia Clinica per la Sperimentazione dei Farmaci, Pisa, Pisa
  - Centro di Ricerche Cliniche di Verona Srl. Policlinico G.B.Rossi, Verona, Verona
- Poland (2):
  - Gabinet Stomatologiczny Andrzej Wojtowicz AW Clinic, Warsaw, Masovian Voivodeship
  - Dental Service spólka jawna, Warsaw, Masovian Voivodeship
- Spain (6):
  - Hospital Médico Quirúrgico de Conxo, Santiago de Compostela, A Coruña
  - Facultad de Odontología. Departamento de Cirugía Bucal y Maxilofacial, University of Barcelona - Bellvitge Institute for Biomedical Research (IDIBELL), L'Hospitalet de Llobregat, Barcelona
  - Universidad Complutense de Madrid, Madrid, Madrid
  - Departamento de Estomatología, Facultad de Odontología. Universidad de Sevilla, Seville, Sevilla
  - Departament d'Estomatologia, Clínica Odontològica, Universidad de Valencia - Fundació Lluís Alcanyís, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
- United Kingdom (3):
  - The School of Dentistry, College of Medical and Dental Sciences, University of Birmingham, Birmingham, England
  - University Dental School Manchester, Manchester, England
  - University Dental Hospital, Cardiff, Wales

REFERENCES:
- [Derived] Moore RA, Gay-Escoda C, Figueiredo R, Toth-Bagi Z, Dietrich T, Milleri S, Torres-Lagares D, Hill CM, Garcia-Garcia A, Coulthard P, Wojtowicz A, Matenko D, Penarrocha-Diago M, Cuadripani S, Piza-Vallespir B, Guerrero-Bayon C, Bertolotti M, Contini MP, Scartoni S, Nizzardo A, Capriati A, Maggi CA. Dexketoprofen/tramadol: randomised double-blind trial and confirmation of empirical theory of combination analgesics in acute pain. J Headache Pain. 2015;16:541. doi: 10.1186/s10194-015-0541-5. Epub 2015 Jun 27. PMID 26123824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in (screening) 23 Feb 2011, last patient out 14 Oct 2011. At 16 study centres in 6 European countries (Germany, Italy, Hungary, Poland, Spain and United Kingdom).
Pre-assignment Details: The trial encompassed 3 visits: 1-Screening; 2-Dental surgery (patients who have moderate to severe pain afterwards were randomised and received study drug); 3-End of study. Overall, 745 patients were enrolled (screened), of them 611 were randomized to receive the study drug and therefore considered as started.
Groups:
- DKP-TRIS 12.5mg - TRAM.HCl 37.5mg: DKP-TRIS 12.5mg - TRAM.HCl 37.5mg oral film-coated tablet, once
- DKP-TRIS 12.5mg - TRAM.HCl 75mg: DKP-TRIS 12.5mg - TRAM.HCl 75mg oral film-coated tablet, once
- DKP-TRIS 25mg - TRAM.HCl 37.5mg: DKP-TRIS 25mg - TRAM.HCl 37.5mg oral film-coated tablet, once
- DKP-TRIS 25mg - TRAM.HCl 75mg: DKP-TRIS 25mg - TRAM.HCl 75mg oral film-coated tablet, once
- DKP-TRIS 12.5mg: DKP-TRIS 12.5mg oral film-coated tablet, once
- DKP-TRIS 25mg: DKP-TRIS 25mg oral film-coated tablet, once
- TRAM.HCl 37.5mg: TRAM.HCl 37.5mg oral film-coated tablet, once
- TRAM.HCl 75mg: TRAM.HCl 75mg oral film-coated tablet, once
- Ibuprofen 400mg: Ibuprofen 400mg oral film-coated tablet, once
- Placebo: Placebo oral film-coated tablet, once
Period: Overall Study
Arm/Group | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg | DKP-TRIS 12.5mg - TRAM.HCl 75mg | DKP-TRIS 25mg - TRAM.HCl 37.5mg | DKP-TRIS 25mg - TRAM.HCl 75mg | DKP-TRIS 12.5mg | DKP-TRIS 25mg | TRAM.HCl 37.5mg | TRAM.HCl 75mg | Ibuprofen 400mg | Placebo
Started | 61 | 63 | 63 | 61 | 60 | 61 | 59 | 60 | 61 | 62
Safety Population | 61 | 63 | 63 | 61 | 60 | 61 | 59 | 60 | 61 | 62
ITT (>= 1 Assessment Post Randomization) | 60 | 62 | 63 | 61 | 60 | 60 | 59 | 59 | 60 | 62
Completed | 61 | 62 | 62 | 60 | 60 | 61 | 58 | 60 | 61 | 62
Not Completed | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Electronic data capture failure | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg | DKP-TRIS 12.5mg - TRAM.HCl 75mg | DKP-TRIS 25mg - TRAM.HCl 37.5mg | DKP-TRIS 25mg - TRAM.HCl 75mg | DKP-TRIS 12.5mg | DKP-TRIS 25mg | TRAM.HCl 37.5mg | TRAM.HCl 75mg | Ibuprofen 400mg | Placebo | Total
Number analyzed (Participants) | 61 | 63 | 63 | 61 | 60 | 61 | 59 | 60 | 61 | 62 | 611
Age Continuous [Mean (Standard Deviation); unit: years] | 28.6 (7.64) | 26.9 (7.62) | 26.3 (7.33) | 27.3 (7.55) | 27.0 (9.85) | 26.9 (6.94) | 25.5 (7.15) | 27.8 (7.99) | 26.6 (6.48) | 26.1 (6.64) | 26.9 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 39 | 36 | 34 | 36 | 44 | 38 | 28 | 41 | 33 | 364
  Male | 26 | 24 | 27 | 27 | 24 | 17 | 21 | 32 | 20 | 29 | 247
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (measured in kg/m^2)
  kg/m^2 | 23.7 (3.39) | 24.1 (3.69) | 23.0 (2.87) | 23.2 (3.19) | 23.6 (3.20) | 23.5 (3.30) | 23.0 (3.19) | 24.2 (3.08) | 22.4 (3.04) | 22.7 (2.80) | 23.3 (3.21)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving at Least 50 % of the Theoretical Maximum Total Pain Relief Score at 6 Hours Post-dosing.
Description: Pain relief is measured by a verbal rating scale (ranging from 0=none to 4=complete). Theoretical maximum TOTPAR at 6 hours is calculated by summing up the maximum score of analgesia which the patient can attribute at defined time points along 6 hour (maxTOTPAR6h= 24). Unit of measure is %
Time Frame: 6 hours
Population: ITT (intention to treat) population which was defined as all patients who have taken the study treatment and have at least 1 post-dose assessment
Measure: Number; unit: percentage of patients
Arm/Group | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg | DKP-TRIS 12.5mg - TRAM.HCl 75mg | DKP-TRIS 25mg - TRAM.HCl 37.5mg | DKP-TRIS 25mg - TRAM.HCl 75mg | DKP-TRIS 12.5mg | DKP-TRIS 25mg | TRAM.HCl 37.5mg | TRAM.HCl 75mg | Ibuprofen 400mg | Placebo
Number analyzed (Participants) | 60 | 62 | 63 | 61 | 60 | 60 | 59 | 59 | 60 | 62
percentage of patients | 36.7 | 59.7 | 55.6 | 72.1 | 26.7 | 55.0 | 10.2 | 25.4 | 45.0 | 9.7

2. Secondary Outcome: Percentage of Patients Achieving at Least 50 % of the Theoretical Maximum Total Pain Relief Score at 4, 8 and 12 Hours Post-dosing.
Description: Pain relief is measured by a verbal rating scale (ranging from 0=none to 4=complete). Theoretical maximum TOTPAR at 6 hours is calculated by summing up the maximum score of analgesia which the patient can attribute at defined time points along 4, 8 and 12 hours(maxTOTPAR4h= 16, maxTOTPAR8h= 32 and maxTOTPAR12h= 48, respectively) Unit of measure is %
Time Frame: 4, 8 and 12 hours
Population: as for outcome 1
Measure: Number; unit: percentage of patient
Arm/Group | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg | DKP-TRIS 12.5mg - TRAM.HCl 75mg | DKP-TRIS 25mg - TRAM.HCl 37.5mg | DKP-TRIS 25mg - TRAM.HCl 75mg | DKP-TRIS 12.5mg | DKP-TRIS 25mg | TRAM.HCl 37.5mg | TRAM.HCl 75mg | Ibuprofen 400mg | Placebo
Number analyzed (Participants) | 60 | 62 | 63 | 61 | 60 | 60 | 59 | 59 | 60 | 62
percentage of patient
  at 4 hours post-dose | 63.3 | 72.6 | 65.1 | 78.7 | 40.0 | 65.0 | 11.9 | 23.7 | 56.7 | 6.5
  at 8 hours post-dose | 21.7 | 48.4 | 44.4 | 54.1 | 16.7 | 31.7 | 6.8 | 20.3 | 33.3 | 6.5
  at 12 hours post-dose | 11.7 | 35.5 | 28.6 | 37.7 | 10.0 | 13.3 | 5.1 | 15.3 | 25.0 | 6.5

3. Secondary Outcome: Percentage of Patients Using Rescue Medication at 6 Hours
Description: Percentage of patients using rescue medication at 6 hours post-dosing.
Time Frame: Baseline to 6 hours
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg | DKP-TRIS 12.5mg - TRAM.HCl 75mg | DKP-TRIS 25mg - TRAM.HCl 37.5mg | DKP-TRIS 25mg - TRAM.HCl 75mg | DKP-TRIS 12.5mg | DKP-TRIS 25mg | TRAM.HCl 37.5mg | TRAM.HCl 75mg | Ibuprofen 400mg | Placebo
Number analyzed (Participants) | 60 | 62 | 63 | 61 | 60 | 60 | 59 | 59 | 60 | 62
percentage of patients | 66.7 | 46.8 | 39.7 | 37.7 | 65.0 | 53.3 | 69.5 | 64.4 | 48.3 | 72.6

ADVERSE EVENTS:
Time Frame: 10 ± 3 days
Description: Analyzed for the Safety population (all patients who received study treatment)
Arm/Group | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg | DKP-TRIS 12.5mg - TRAM.HCl 75mg | DKP-TRIS 25mg - TRAM.HCl 37.5mg | DKP-TRIS 25mg - TRAM.HCl 75mg | DKP-TRIS 12.5mg | DKP-TRIS 25mg | TRAM.HCl 37.5mg | TRAM.HCl 75mg | Ibuprofen 400mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/63 | 0/63 | 0/61 | 0/60 | 0/61 | 0/59 | 1/60 | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 7/61 | 9/63 | 6/63 | 10/61 | 2/60 | 4/61 | 5/59 | 14/60 | 5/61 | 1/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg (N=61) | DKP-TRIS 12.5mg - TRAM.HCl 75mg (N=63) | DKP-TRIS 25mg - TRAM.HCl 37.5mg (N=63) | DKP-TRIS 25mg - TRAM.HCl 75mg (N=61) | DKP-TRIS 12.5mg (N=60) | DKP-TRIS 25mg (N=61) | TRAM.HCl 37.5mg (N=59) | TRAM.HCl 75mg (N=60) | Ibuprofen 400mg (N=61) | Placebo (N=62)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DKP-TRIS 12.5mg - TRAM.HCl 37.5mg (N=61) | DKP-TRIS 12.5mg - TRAM.HCl 75mg (N=63) | DKP-TRIS 25mg - TRAM.HCl 37.5mg (N=63) | DKP-TRIS 25mg - TRAM.HCl 75mg (N=61) | DKP-TRIS 12.5mg (N=60) | DKP-TRIS 25mg (N=61) | TRAM.HCl 37.5mg (N=59) | TRAM.HCl 75mg (N=60) | Ibuprofen 400mg (N=61) | Placebo (N=62)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 1 (2) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (4) | 3 (3) | 5 (6) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the investigator will allow the Sponsor at least 60 days time to review and comment upon the publication manuscript. It is agreed, that the results of the study will not be submitted for presentation, abstract, poster exhibition, or publication by the investigator until the Sponsor has reviewed/commented and agreed to any publication.